CLINICAL TRIAL: NCT00305526
Title: Resynchronisation and Beta-Blocker European Trial
Brief Title: REBEAT Resynchronisation and Beta-Blocker European Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of enrolment
Sponsor: Guidant Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REBEAT 1.5
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: Contak Renewal (CRT-D)

SUMMARY:
This protocol will evaluate the effect of cardiac resynchronization therapy (CRT) combined with beta-blocker therapy in patients with symptomatic heart failure in whom beta-blocker therapy was either not tolerated or could not be up titrated to optimal doses before CRT. Cardiac resynchronization therapy will be combined with automatic implantable cardioverter defibrillator (AICD, CRT-D) as it has been shown to be associated with an improvement in prognosis in the patients with left ventricular systolic dysfunction and heart failure.

DETAILED DESCRIPTION:
The purpose of this investigation is to evaluate the effect of CRT combined with beta-blocker therapy in patients with symptomatic heart failure in whom beta-blocker therapy was either not tolerated or could not be up-titrated to optimal doses before CRT.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure and indication for cardiac resynchronization therapy (CRT), Hemodynamic stability with documented intolerance to beta-blocker therapy or treatment with beta-blocking agents at sub-optimal dosages (<25% of optimal dosage).

Exclusion Criteria:

* chronic atrial fibrillation; indications for permanent antibradycardia pacing; mechanical tricuspid valve; Severe aortic stenosis or other primary valve disease causing cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2006-04; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
LVEF changes between baseline and 6 months measured by Echocardiography

SECONDARY OUTCOMES:
increase % of patients with successful uptitration for Betablockers, reduce all cause hospitalizations and all cause mortality, reduce all cause mortality and heart failure hospitalizations, reduce all cause mortality and cardiovascular hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curnis, MD, Principal Investigator — Spedali Civili di Brescia, Brescia, Italy
Locations (3):
- Italy (2):
  - Spedali Civili di Brescia, Brescia
  - Istituto clinico Humanitas, Milan
- Cardiocentro Ticino, Lugano, Switzerland